CLINICAL TRIAL: NCT03194750
Title: Ultrasound Assessment of Volume in Patients on Continuous Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eric Judd, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: F160407004
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Volume Overload; Kidney Failure; Respiratory Failure
MeSH Terms: conditions — Edema; Renal Insufficiency; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Share Data (Experimental)
  Interventions: Other: Share ultrasound measurement of IVC collapsibility to Nephrology Attending
- Do Not Share Data (Active Comparator)
  Interventions: Other: Do not share ultrasound measurement of IVC collapsibility to Nephrology Attending

INTERVENTIONS:
Other: Share ultrasound measurement of IVC collapsibility to Nephrology Attending — Nephrology attending will be provided with the respiratory variability of IVC diameter as a percent, in addition to a predefined cutoff for responsiveness to volume resuscitation of < 12%. The information will be provided before rounds and before the attending sets the fluid removal goals on dialysis for that day.
  Arms: Share Data
Other: Do not share ultrasound measurement of IVC collapsibility to Nephrology Attending — Respiratory variability of IVC diameter will be measured, but the measurement result will not be shared with the treating team.
  Arms: Do Not Share Data

SUMMARY:
Renal failure and resuscitation measures in critically ill patients can result in fluid overload. Fluid overload in renal failure patients can cause harmful effects like pulmonary edema, anasarca and congestive cardiac failure exacerbations among other complications. These have been associated with increased time on the ventilator, increased length of stay in the ICU, and higher overall mortality for patients requiring dialysis in the ICU.

The current standard of care for adjusting fluid removal rates in patients on continuous renal replacement therapy relies on clinical judgement. Clinicians take into account factors like the patient's condition, vasopressor requirements, kidney function, total intake and outputs, vital signs, and physical examination findings when making daily changes to fluid removal rates on dialysis machines. Such assessment is highly subjective and can be imprecise/inaccurate leading to hypotension and hemodynamic instability in a critically ill patient.

Use of conventional ultrasound by physicians to assess volume status using compressibility of the inferior vena cava has been shown to be a reliable predictor of volume status and can help guide therapy. Such use makes bedside volume assessment a non-invasive, rapid, repeatable point of care tool that can provide objective data to guide fluid removal determine velocity of fluid removal and help identify patients at risk of hypotension and hemodynamic instability during the process of fluid removal. Apart from rare possible local allergic reactions to ultrasound jelly and transient local discomfort, the disadvantages are minimal. Ultrasonography has been considered a safe imaging modality. This protocol will measure inferior vena cava compressibility using the General Electric VScan with Dual Probe, which has FDA approval for abdominal and vascular imaging in humans.

DETAILED DESCRIPTION:
The study consists of gathering patient data from the chart and performing ultrasound measurements of inferior vena cava compressibility at the start of continuous renal replacement therapy (CRRT) in patients on the mechanical ventilator in the ICU. Ultrasound measurements on the abdomen, as well as recording of clinical data like intake/output, weight, pulse pressure variability, vasopressor requirement, nutrition requirement, ventilator settings, CRRT settings, and certain laboratory data will be performed at the start of the study and then daily for the next 3 days. On the 3rd day, 50 mL of dialysis waste fluid will be collected and stored for future analysis.

At the start of the study, participants will be randomized to two groups. Study activities are identical between the two groups and both groups receive ultrasound measurements on the abdomen. However, in one group the attending nephrologist on the Acute Consult service will be provided with inferior vena cava compressibility measurement information each day before the start of rounds. Randomization will follow a predefined schedule, known only to the research coordinator, Laura Latta. At no time will the attending physicians receive the ultrasound measurements for the group randomized to not have their data shared.

In addition, the resident, fellow, and attending on the Acute Consult service will be asked to assess the volume status of each participant at the start of the study and then daily for next 3 days. The volume assessment will consist of answering the following question, "Would you recommend fluid removal in this patient today (Yes/No/Unsure)?" The question will be asked verbally by Dr. Narasimha Krishna. Each individual's level of training (post-graduation year) and the response will be recorded. Individual names will not be recorded and responses will not be shared with the attending. Responses to this question are not anticipated to affect management of the participant.

During the follow up phase, the electronic medical records will be checked at day 7 and day 30 to determine if the participant is still in the intensive care unit, is still on the ventilator, or is still alive, or still in the hospital. Both groups will have the same follow up time.

Primary outcome measures include: 1) Time to extubation; 2) Length of ICU stay; 3) Length of hospital stay; and 4) 30 day mortality.

Secondary outcome measures include: 1) Difference in net fluid removal by CRRT at day 3 between the 2 groups; 2) Agreement between volume assessment and inferior vena cava compressibility by level of training.

ELIGIBILITY:
Inclusion Criteria:

* Acute kidney injury requiring initiation of continuous renal replacement therapy
* Respiratory failure requiring mechanical ventilation

Exclusion Criteria:

* cirrhosis of liver
* pregnant woman
* abdominal surgery interfering with placement of ultrasound probe
* end-stage kidney disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Time to extubation | Start of study to up to 30 days
  Length of time the participant is intubated from the start of the study up until the 30 day chart follow up.
Length of ICU stay | Start of study to up to 30 days
  Length of time the participant remains in the ICU from the start of the study up until chart follow up at 30 days.
Length of hospital stay | Start of study to up to 30 days
  Length of time the participant remains in the hospital up until the 30 day chart follow up.
30 day mortality | Start of study to day 30

SECONDARY OUTCOMES:
Difference in net fluid removal by CRRT at day 3 | Start of study to day 3
  As measured by documented total intake and output
Agreement between volume assessment and inferior vena cava collapsibility by level of training. | Start of study to day 3
  As measured by a kappa statistic between a yes/no question and a predefined IVC collapsibility threshold for fluid removal.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Judd, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB University Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No